CLINICAL TRIAL: NCT02319811
Title: Meniscus Transplantation in Symptomatic Patients Under Fifty Years of Age: Survivorship Analysis
Brief Title: Cryopreserved Human Meniscus Transplantation
Status: Completed | Type: Observational
Sponsor: Cincinnati Sportsmedicine Research and Education Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MenisCryo-001
Record Dates: First submitted 2014-12-10; First posted 2014-12-18 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cryopreserved meniscus transplant: Intervention: Lateral or medial cryopreserved meniscus transplant implanted into appropriately indicated patients.
  Interventions: Procedure: Cryopreserved meniscus transplants

INTERVENTIONS:
Procedure: Cryopreserved meniscus transplants — Lateral or medial cryopreserved meniscus transplants implanted into appropriately indicated patients.

SUMMARY:
The purpose of this study is to determine the long-term survivorship and clinical outcomes of all cryopreserved meniscus transplants performed by Dr. Frank Noyes.

DETAILED DESCRIPTION:
All patients receiving cryopreserved meniscus transplants will be followed at 1, 2, 5, 10, and 15 years postoperatively. Study examination will include comprehensive knee examination by Dr. Noyes, x-rays, and potentially MRI. Patients will complete the following forms of the Cincinnati Knee Rating System: Symptom Rating Form, Sports Activity and Function Form, and Occupational Rating Form. All patient identification will be kept confidential. Patient data will be entered into the Knee Registry database according to their unique study number by the clinical research assistant.

ELIGIBILITY:
Inclusion Criteria:

* Patient post-meniscectomy
* Patient symptomatic with activities
* Patient has early articular cartilage degeneration in affected tibiofemoral compartment
* Patient understands goals of operation, willing to undergo lengthy rehabilitation

Exclusion Criteria:

* Patient has no symptoms with activities
* Patient has advanced degeneration in affected tibiofemoral compartment or other compartments
* Patient is obese (BMI > 30)
* Patient has uncorrected lower limb axial malalignment or knee ligament deficiency
* Patient has active infection
* Patient has pre-existing knee arthrofibrosis or lower limb muscular atrophy
* Patient has symptomatic patellofemoral articular cartilage deterioration
* Patient is unwilling to undergo lengthy rehabilitation after surgery

Ages: 14 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Minimum age: 14 Years Maximum age: 49 Years Gender: Both Accepts Healthy Volunteers: No Patients post-meniscectomy, symptomatic with activities, early cartilage degeneration in affected tibiofemoral compartment.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 1995-11; Primary Completion 2014-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Survivorship analysis | 15 years postoperatively

SECONDARY OUTCOMES:
Cincinnati Knee Rating System | 15 years postoperatively
  The following factors will be scored according to the validated Cincinnati Knee Rating System: pain, swelling, giving-way, walking, stair-climbing, squatting, running, jumping, pivoting, sports activity level, occupational level, patient perception of the knee condition.
International Knee Documentations Committee | 15 years postoperatively
  The validated IKDC overall evaluation form will be used to rate knee function.

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Noyes, M.D., Principal Investigator — President, Noyes Knee Institute

IPD SHARING:
Plan to Share IPD: Yes
Published results in Journal of Bone and Joint Surgery, 2015 and American Journal of Sports Medicine 2016